CLINICAL TRIAL: NCT03612700
Title: Presence of Cyclopropane Fatty Acids (CPFA) in Human Plasma After CPFA-rich Diet
Brief Title: Presence of Cyclopropane Fatty Acids (CPFA) in Human Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Daniele Del Rio, Professor, University of Parma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DDR-CPFA
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Biological Availability
Keywords: Cyclopropane fatty acids; GC-MS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPFA-rich diet (Experimental): Free living diet controlled in CPFA intake
  Interventions: Other: CPFA-rich foods

INTERVENTIONS:
Other: CPFA-rich foods — Daily consumption of Grana Padano cheese (50 g) and whole milk (250 mL) for 3 weeks.

SUMMARY:
Fatty acids containing a cyclopropane ring in their structure (CPFA) have been found in plants, fungi, a wide variety of bacteria and recently detected in dairy products and bovine meat. Little is known about CPFA in mammals, especially in human tissues. This work aims at investigating the presence of CPFA in plasma of humans after a regular consumption of CPFA from milk and cheese. A free living diet controlled in CPFA, mainly deriving from Grana Padano cheese and whole milk containing CPFA, will be consumed by 10 healthy normal weight volunteers for three weeks, after one week of dairy products and bovine meat restricted diet. Plasma of volunteers will be collected at 8 different timepoints for lipid extraction, CPFA identification and quantification by GC-MS. A preliminary pilot in vivo acute study (involving only 1 subject) will be performed for investigating the post-prandial response curve of CPFA after a portion of Grana Padano cheese.

DETAILED DESCRIPTION:
Cyclopropane fatty acids (CPFA), as cis-9,10- methyleneoctadecanoic and cis- 11,12- methyleneoctadecanoic acids, are unusual alicyclic fatty acids which occur in plants, fungi, or microorganisms both Gram-negative and Gram-positive as well as protozoa and Myriapoda. Some papers suggest that cyclopropane fatty acids are involved in the bacterial pathogenesis of infections and in the resistance of some bacterial strains as Lactobacillus sp., Escherichia Coli, Salmonella enterica, Staphilococcus aureus and Pseudomonas to different environmental stresses such as temperature changes, high osmolarity, solvents, acid pH and others as the presence of antibiotics or heavy metals in the culture medium. However, little is documented about the presence of CPFA in mammals. Recently, they were detected in milk and several dairy products, in bovine meat, in fish and in mushrooms. Our previous results showed that the most important food sources of CPFA were dairy products (mainly Grana Padano cheese) and bovine meat reaching concentration of 1g/kg order, while food processing, manufacturing, seasoning steps, fermentation as well as cooking did not affect CPFA content in the analyzed food matrices. Furthermore, CPFA intake from these foodstuffs should be considered dietary relevant in view of a possible physiological effect.

Actually, CPFA (mainly cyclopropaneoctanoic acid 2-hexyl) have been recently identified in both human serum and adipose tissue, suggesting that these fatty acids are efficiently absorbed and may play a physiological role in the human body.

Moreover, fatty acids containing cyclopropane rings have been reported to exert biological effects on lipid metabolism, kidney function, inflammation, and enzymes activity as cyclooxygenase and stearoyl-CoA desaturase. Previous results suggested that the synthesis of CPFA in microorganisms and in plants is regulated by the expression of CPFA synthase, which catalyse the addition of the methylene group from S-adenosylmethionine to double bond of the unsaturated fatty acids precursor. However, this enzyme has still not been identified in animals and humans. To the best of our knowledge, no information is present in literature about the fate of CPFA within the human body, and a thorough investigation of how CPFA can be metabolised and accumulate in humans is needed.

The aim of this investigation is to determine CPFA presence in human plasma after a CPFA-rich diet (with controlled intake of Grana Padano cheese and whole milk containing CPFA). Plasma of the volunteers will be collected at eight different timepoints for lipid extraction, CPFA identification and quantification by GC-MS. A preliminary pilot in vivo acute study will be performed (involving only 1 subject) for investigating the post-prandial response curve of CPFA after a portion of Grana Padano cheese.

ELIGIBILITY:
Inclusion Criteria:

- BMI 19-29 (kg/m2)

Exclusion Criteria:

* pregnancy and lactation
* gastrointestinal disorders
* metabolic diseases
* drugs and food supplements interfering with lipid metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
CPFA plasmatic concentration | Fasting CPFA plasma concentration [time -7 days, time 0 (after 1 week of CPFA restricted diet), time 3, 6, 9, 12, 15, 18 days]
  Fasting concentration of CPFA

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Del Rio, Professor, Principal Investigator — Department of Food and Drugs; Augusta Caligiani, Professor, Principal Investigator — Department of Food and Drugs
Locations (1):
- Department of Food and Drugs, University of Parma, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore BS, Floss HG. Biosynthesis of Cyclic Fatty Acids Containing Cyclopropyl-, Cyclopentyl-, Cyclohexyl-, and Cycloheptyl-rings. Reference Module in Chemistry, Molecular Sciences, and Chemical Engineering, from Comprehensive Natural Products Chemistry 1:61-82, 1999
- [Background] Montanari C, Sado Kamdem SL, Serrazanetti DI, Etoa FX, Guerzoni ME. Synthesis of cyclopropane fatty acids in Lactobacillus helveticus and Lactobacillus sanfranciscensis and their cellular fatty acids changes following short term acid and cold stresses. Food Microbiol. 2010 Jun;27(4):493-502. doi: 10.1016/j.fm.2009.12.003. Epub 2010 Jan 6. PMID 20417398
- [Background] Poger D, Mark AE. A ring to rule them all: the effect of cyclopropane Fatty acids on the fluidity of lipid bilayers. J Phys Chem B. 2015 Apr 30;119(17):5487-95. doi: 10.1021/acs.jpcb.5b00958. Epub 2015 Apr 16. PMID 25804677
- [Background] Marseglia A, Caligiani A, Comino L, Righi F, Quarantelli A, Palla G. Cyclopropyl and omega-cyclohexyl fatty acids as quality markers of cow milk and cheese. Food Chem. 2013 Oct 15;140(4):711-6. doi: 10.1016/j.foodchem.2013.01.029. Epub 2013 Jan 23. PMID 23692757
- [Background] Caligiani A, Marseglia A, Palla G. An overview on the presence of cyclopropane fatty acids in milk and dairy products. J Agric Food Chem. 2014 Aug 6;62(31):7828-32. doi: 10.1021/jf4057204. Epub 2014 Jul 24. PMID 25033416
- [Background] Sledzinski T, Mika A, Stepnowski P, Proczko-Markuszewska M, Kaska L, Stefaniak T, Swierczynski J. Identification of cyclopropaneoctanoic acid 2-hexyl in human adipose tissue and serum. Lipids. 2013 Aug;48(8):839-48. doi: 10.1007/s11745-013-3806-2. Epub 2013 Jun 11. PMID 23754307
- [Background] Bichi E, Toral PG, Hervas G, Frutos P, Gomez-Cortes P, Juarez M, de la Fuente MA. Inhibition of ∆9-desaturase activity with sterculic acid: effect on the endogenous synthesis of cis-9 18:1 and cis-9, trans-11 18:2 in dairy sheep. J Dairy Sci. 2012 Sep;95(9):5242-5252. doi: 10.3168/jds.2012-5349. PMID 22916929
- [Background] Jones SE, Whitehead K, Saulnier D, Thomas CM, Versalovic J, Britton RA. Cyclopropane fatty acid synthase mutants of probiotic human-derived Lactobacillus reuteri are defective in TNF inhibition. Gut Microbes. 2011 Mar-Apr;2(2):69-79. doi: 10.4161/gmic.2.2.15282. Epub 2011 Mar 1. PMID 21637024
- [Background] Kadegowda AK, Burns TA, Pratt SL, Duckett SK. Inhibition of stearoyl-CoA desaturase 1 reduces lipogenesis in primary bovine adipocytes. Lipids. 2013 Oct;48(10):967-76. doi: 10.1007/s11745-013-3823-1. Epub 2013 Aug 9. PMID 23929455
- [Background] Mika A, Stepnowski P, Chmielewski M, Malgorzewicz S, Kaska L, Proczko M, Ratnicki-Sklucki K, Sledzinski M, Sledzinski T. Increased Serum Level of Cyclopropaneoctanoic Acid 2-Hexyl in Patients with Hypertriglyceridemia-Related Disorders. Lipids. 2016 Jul;51(7):867-73. doi: 10.1007/s11745-016-4141-1. Epub 2016 Mar 22. PMID 27003900
- [Background] Schneider AC, Beguin P, Bourez S, Perfield JW 2nd, Mignolet E, Debier C, Schneider YJ, Larondelle Y. Conversion of t11t13 CLA into c9t11 CLA in Caco-2 cells and inhibition by sterculic oil. PLoS One. 2012;7(3):e32824. doi: 10.1371/journal.pone.0032824. Epub 2012 Mar 12. PMID 22427892
- [Background] Grogan DW, Cronan JE Jr. Cyclopropane ring formation in membrane lipids of bacteria. Microbiol Mol Biol Rev. 1997 Dec;61(4):429-41. doi: 10.1128/mmbr.61.4.429-441.1997. PMID 9409147
- [Background] WOOD R, REISER R. CYCLOPROPANE FATTY ACID METABOLISM: PHYSICAL AND CHEMICAL IDENTIFICATION OF PROPANE RING METABOLIC PRODUCTS IN THE ADIPOSE TISSUE. J Am Oil Chem Soc. 1965 Apr;42:315-20. doi: 10.1007/BF02540137. No abstract available. PMID 14279117
- [Background] Wessjohann LA, Brandt W, Thiemann T. Biosynthesis and metabolism of cyclopropane rings in natural compounds. Chem Rev. 2003 Apr;103(4):1625-48. doi: 10.1021/cr0100188. No abstract available. PMID 12683792
- [Background] Kim BH, Kim S, Kim HG, Lee J, Lee IS, Park YK. The formation of cyclopropane fatty acids in Salmonella enterica serovar Typhimurium. Microbiology (Reading). 2005 Jan;151(Pt 1):209-218. doi: 10.1099/mic.0.27265-0. PMID 15632439
- [Background] Lolli V, Marseglia A, Palla G, Zanardi E, Caligiani A. Determination of Cyclopropane Fatty Acids in Food of Animal Origin by 1H NMR. J Anal Methods Chem. 2018 Apr 1;2018:8034042. doi: 10.1155/2018/8034042. eCollection 2018. PMID 29805838
- [Result] Bao X, Katz S, Pollard M, Ohlrogge J. Carbocyclic fatty acids in plants: biochemical and molecular genetic characterization of cyclopropane fatty acid synthesis of Sterculiafoetida. Proc Natl Acad Sci U S A. 2002 May 14;99(10):7172-7. doi: 10.1073/pnas.092152999. Epub 2002 May 7. PMID 11997456